CLINICAL TRIAL: NCT06346808
Title: Oncolytic Virus Plus Anti-PD1 and Chemotherapy as Preoperative Therapy for Patients With Borderline Resectable and Locally Advanced Pancreatic Cancer
Brief Title: Oncolytic Virus Plus Anti-PD1 and Chemotherapy as Preoperative Therapy for Patients With BRPC/LAPC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDAC-OV
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Oncolytic virus; immunotherapy; Preoperative therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic virus Plus Anti-PD1 and Chemotherapy (Experimental): Oncolytic virus d1 ;Camrelizumab 200mg, d2+AG(Gemcitabine d2/9+Capecitabine d2-d15),q3w；up to 4 cycles;
  Interventions: Drug: Oncolytic virus Plus Anti-PD1 and Chemotherapy

INTERVENTIONS:
Drug: Oncolytic virus Plus Anti-PD1 and Chemotherapy — Oncolytic virus，Camrelizumab ，AG（Gemcitabine +Capecitabine ）

SUMMARY:
The aim of this single center, single arm and prospective study is to explore the safety and efficacy of Oncolytic virus Plus Anti-PD1 and Chemotherapy as Preoperative therapy for Patients with Borderline Resectable and Locally Advanced Pancreatic Cancer

ELIGIBILITY:
Inclusion Criteria:

- Age ≥18 years and age ≤75 years. ECOG score 0-1. Patients with Borderline Resectable and Locally Advanced Pancreatic Cancer

Adequate bone marrow and organ function:

Patients of childbearing potential must take appropriate precautions prior to enrollment and during the study.

Signed informed consent. Ability to comply with the study protocol and follow-up.

Exclusion Criteria:

1. Received antitumor chemotherapy, radiation therapy, and immunotherapy prior to first treatment.
2. Patients with comorbid severe pancreatic portal hypertension, which may cause a higher risk of bleeding with subsequent injection therapy;
3. Patients with prior or concomitant history of other tumors (except basal cell carcinoma of the skin, cervical cancer in situ).
4. Serious uncontrolled medical conditions that may interfere with the subject's ability to receive treatment as specified in the protocol, including, but not limited to, positive HIV test, active tuberculosis, and DNA copy number of HBV >103/ml;
5. Uncontrollable comorbidities, including, but not limited to, active bacterial, viral, tuberculosis, or fungal infection, symptomatic congestive heart failure, unstable angina, and cardiac arrhythmia.
6. Patients with autoimmune disease or immunodeficiency treated with immunosuppressive drugs;
7. Pregnant or lactating women;
8. Those who may be allergic to the study drug or any of its excipients;
9. Preoperative ultrasound evaluation of patients with small tumor size, location near or behind major blood vessels, and various other factors that may result in a low success rate of intra-tumoral viral injection under ultrasound and a high rate of post-injection complications;
10. Substance abuse or those who are unable to undergo immunization or lysosomal viral therapy due to clinical, psychological, or social factors.
11. Any uncertainty that affects patient safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year
  Defined by treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
R0 resection rate | 6 months
  defined as complete resection without any macroscopic or microscopic evidence of lesion at the lateral and deep tissue margins
ORR | 6 months
  The incidence of CR (complete remission) and PR (partial remission)

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No